CLINICAL TRIAL: NCT07168876
Title: Clinical Validation Cross-sectional Study for Colorectal Cancer Assessment Using Delta-HLD Technology (CLIMBED)
Brief Title: Colon Cancer Liquid Biopsy Investigation of Methylation-based Biomarkers Evaluation Using Delta-HLD (CLIMBED)
Acronym: CLIMBED
Status: Recruiting | Type: Observational
Sponsor: Epiliquid Holding, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: CRC-CV; RENIS IS004624 (Other: Epiliquid Holding, Inc)
Record Dates: First submitted 2025-09-04; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2024-09

CONDITIONS: Colorectal Cancer (CRC)
Keywords: Colorectal cancer; Epigenetics; Liquid biopsy; cfDNA; Biomarker; Methylarion; PCR
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Plasma samples will be collected and retained for analysis. Circulating cell-free DNA (cfDNA) will be extracted from plasma and stored for future validation studies. No other sample types will be retained.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cases: Average-risk population undergoing colorectal cancer screening colonoscopy

SUMMARY:
CLIMBED (Colon cancer Liquid biopsy Investigation of Methylation-based Biomarkers Evaluation using Delta-HLD) is a non-randomized, observational, cross-sectional clinical validation study designed to assess the performance of Delta-HLD, Epiliquid's proprietary liquid biopsy technology, for colorectal cancer (CRC) detection. The study will evaluate the test performance in an average-risk population for CRC undergoing screening colonoscopy, which will serve as the gold standard reference.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is one of the most common cancers worldwide and among the leading causes of cancer-related mortality. Early detection substantially improves survival; however, adherence to existing screening strategies remains suboptimal across different regions. CLIMBED is a non-randomized, observational, cross-sectional clinical validation study designed to assess the performance of Epiliquid's Delta-HLD liquid biopsy technology, which detects methylation-based epigenetic biomarkers in plasma using PCR. The study will enroll 3200 participants between 45 and 75 years of age, representing an average-risk CRC population. All participants will undergo screening colonoscopy, which will serve as the gold standard for comparison. The primary endpoints are sensitivity, specificity, positive predictive value (PPV), and negative predictive value (NPV) of the Delta-HLD technology for CRC detection in cfDNA. Secondary endpoints include the capacity of the test to identify precursor lesions. Statistical analysis will be based on ROC curves and AUC to determine diagnostic performance.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 45-75 years
* Indication of colorectal cancer screening colonoscopy by treating physician

Exclusion Criteria:

* First-degree family history of CRC
* Inflammatory bowel disease (ulcerative colitis, Crohn's disease)
* Other malignancies within 5 years
* Known hereditary CRC syndromes (Lynch, FAP)
* Major trauma, surgery, transfusion in past 30 days
* Current participation in an interventional clinical trial

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Single cohort of adults aged 45 and 75 years, representing an average-risk CRC population, undergoing routine colorectal cancer screening with colonoscopy in Argentina as standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 3200 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of colorectal cancer detection | 18 months
  Sensitivity and specificity of the Delta-HLD test for detection of colorectal cancer
Specificity of advanced neoplasia detection | 36 months
  Specificity of colorectal cancer detection

SECONDARY OUTCOMES:
Accuracy of colorectal cancer precursor lesions detection | 36 months
  Sensitivity and specificity of of colorectal cancer precursor lesions detection
Predictive values | 36 months
  Positive predictive value (PPV) and negative predictive value (NPV) of the Delta-HLD test for CRC detection

CONTACTS AND LOCATIONS:
Overall Officials: Emanuel Campoy, PhD, Study Director — CONICET-National Scientific and Technical Research Council
Locations (1):
- Epiliquid, Mendoza, Mendoza Province, Argentina

IPD SHARING:
Plan to Share IPD: No